CLINICAL TRIAL: NCT02145910
Title: Phase I Study of Vemurafenib Combined With Whole Brain Radiation Therapy (WBRT) or Radiosurgery (SRS) for Melanoma Patients With BRAF Mutation Presented With Brain Metastases
Brief Title: Vemurafenib Combined With Whole Brain Radiation Therapy or Radiosurgery in Patients With BRAF Mutation-Positive Melanoma and Brain Metastases
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never opened to accrual. There is no clinical benefit to patients.
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13P.480; 2013-025 (Other: CCRRC); JT 2960 (Other: JeffTrial Number)
Record Dates: First submitted 2014-05-13; First posted 2014-05-23 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Melanoma; Stage IV Melanoma; Tumors Metastatic to Brain
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — Vemurafenib; Radiosurgery; Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WBRT + Vemurafenib (Experimental): Patients undergo WBRT once daily (QD) for 10 doses
  Interventions: Drug: Vemurafenib; Radiation: Whole-brain radiation therapy (WBRT)
- SRS + Vemurafenib (Experimental): Patients undergo SRS (gamma knife, tomotherapy, cyberknife, or megavoltage LINAC radiation therapy) on day 1
  Interventions: Drug: Vemurafenib; Radiation: Radiosurgery (SRS)

INTERVENTIONS:
Drug: Vemurafenib — Given PO
  Other Names: Zelboraf
Radiation: Whole-brain radiation therapy (WBRT) — Undergo WBRT
  Other Names: WBRT; whole brain radiotherapy; whole-brain radiotherapy
  Arms: WBRT + Vemurafenib
Radiation: Radiosurgery (SRS) — Undergo SRS
  Other Names: Radiation surgery; SRS
  Arms: SRS + Vemurafenib

SUMMARY:
This phase I trial studies the best dose of vemurafenib when combined with whole brain radiation therapy (WBRT) or stereotactic radiosurgery (SRS) in patients with v-raf murine sarcoma viral oncogene homolog B (BRAF) mutation-positive melanoma and brain metastases. Radiation therapy is an effective treatment for patients with brain metastases. Patients with multiple metastases are typically treated with WBRT. For patients with a few metastases, SRS alone can be used. Vemurafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Combining radiation treatment with vemurafenib for melanoma patients with brain metastases may result in improved local control and prolonged survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of vemurafenib when combined with WBRT or SRS and determine a recommended phase II dose of vemurafenib to be used with WBRT or SRS in patients with brain metastases from melanoma.

SECONDARY OBJECTIVES:

I. To determine local control rates of the brain metastases in each arm. II. To determine the rates of developing of new brain metastases in each arm. III. To determine the response of extracranial disease. IV. To determine the overall survival rate and progression free survival rate. V. To determine the safety and tolerability of each arm.

OUTLINE: This is a dose-escalation study of vemurafenib. Patients are assigned to 1 of 2 arms based on the number and size of brain metastasis.

All patients receive vemurafenib orally (PO) twice daily (BID) beginning 3-5 days before the start of radiation therapy and continuing in the absence of disease progression or unacceptable toxicity.

ARM A: Patients undergo WBRT once daily (QD) for 10 doses.

ARM B: Patients undergo SRS (gamma knife, tomotherapy, cyberknife, or megavoltage linear accelerator [LINAC] radiation therapy) on day 1.

After completion of study therapy, patients are followed up on weeks 5 or 7, 9 and 13, and then on months 4, 6, 9, and 12.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histological confirmed melanoma (prior diagnosis okay)
3. BRAFV600 mutation positive (cobas 4800 BRAFV600 mutation test)
4. ECOG performance status 0 or 1
5. Craniotomy resection is allowed (a minimum 2 weeks recovery time from surgery to initiation of protocol therapy)
6. Radiographic evidence of brain metastasis
7. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
8. Adequate organ function:

   1. WBC ≥ 2000/uL
   2. ANC ≥ 1000/uL
   3. Platelets ≥ 75 x 103/uL
   4. Hemoglobin ≥ 9 g/dL (≥ 80 g/L; may be transfused)
   5. Creatinine ≤ 2.0 x ULN OR 24-hour creatinine clearance >= 50 ml/min
   6. AST/ALT ≤ 2.5 x ULN for patients without liver metastasis, ≤ 5 times for liver metastases
   7. Bilirubin ≤ 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
   8. Total serum calcium (corrected for serum albumin) or ionized calcium ≥ lower limit of normal (LLN)
   9. Serum potassium ≥ LLN
   10. Serum sodium ≥ LLN
   11. Serum albumin ≥ LLN or 3g/dl
   12. Patients with any elevated Alkaline Phosphatase due to bone metastases can be enrolled
9. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized. Women of potential child bearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:

   1. Amenorrhea ≥ 12 consecutive months without another cause, or
   2. For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level ≥ 35 mIU/mL.
   3. Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.
   4. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of radiation.

   Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.
10. Specific eligibility criteria for the two arms:

    1. Arm A (WBRT and Vemurafenib):

       * Patients have 5 or more brain metastases, or patients have any brain metastases exceeding the limit for SRS (maximum diameter is > 4 cm).
       * OR Patient has only one brain metastasis and completely resected, the resection cavity is > 5 cm in diameter.
    2. Arm B (SRS and Vemurafenib):

       * Patients have 4 or fewer brain metastases. All the brain metastases are ≤ 4 cm in diameter.
       * Patients have only one brain metastasis and completely resected, the resection cavity is ≤ 5 cm in diameter.
       * OR If a patient is found to have progression of brain metastases that exceed 4 cm in diameter based on the MRI scan on the day of SRS procedure, the patient should be re-assigned to WBRT arm or withdrawn from the study. The study PI should be notified.
       * OR If a patient is found to have progression of brain metastases that exceed 4 lesions based on the MRI scan on the day of the SRS procedure, the patient can either receive SRS to all the lesions (up to 10 lesions), be re-assigned to WBRT arm, or be withdrawn from the study per the treating physician. The study PI should be notified.

Exclusion Criteria:

1. Leptomeningeal involvement
2. Cardiac disease: Congestive heart failure > class II. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
3. Pregnancy or breastfeeding
4. Documented history of cranial hemorrhage
5. Concurrent administration of any anticancer therapies other than those administered in the study
6. Treatment with any cytotoxic, investigational drug, or targeted therapy within 2 weeks prior to the protocol treatment.
7. Craniotomy within 2 weeks of protocol treatment.
8. Prior treatment with other BRAF or MEK inhibitors
9. Patients who had prior brain radiation. However, prior WBRT is allowed in Arm B.
10. QTc > 450 ms
11. Patients have a history of any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated basal or squamous cell carcinoma of skin, superficial bladder cancer or carcinoma in situ of cervix, AJCC (version 7.0) stage 0 or I breast cancer, AJCC (version 7.0) stage I, or II prostate cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of vemurafenib | Up to 1 year
  The last dose studied or the previous dose, based on clinical judgment of the degree of toxicity seen at the last dose.

SECONDARY OUTCOMES:
Proportion with complete response | Up to 1 year
  Estimate through the Kaplan-Meier method and compute associated 95% confidence intervals
Proportion with partial response | Up to 1 year
  Estimate through the Kaplan-Meier method and compute associated 95% confidence intervals
Median survival | Up to 1 year
  Estimate through the Kaplan-Meier method and compute associated 95% confidence intervals
Progression free survival based on Response Evaluation Criteria In Solid Tumors (RECIST) criteria based on the brain MRI and systematic assessment by the treating physician | Up to 1 year
  Will be determined for each arm separately, as well as the entire study patient population
Overall survival | Up to 1 year
  Will be determined for each arm separately, as well as the entire study patient population
Local control rates of brain metastases | Up to 1 year
  Analysis of local control will be done separately in each arm
Rate of developing new brain metastasis | Up to 1 year
  Analysis of rate of developing new brain metastasis will be done separately in each arm
Response of extracranial disease | Up to 1 year
  Will be determined for each arm separately, as well as the entire study patient population

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, PhD, Principal Investigator — Thomas Jefferson University

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org